CLINICAL TRIAL: NCT02286908
Title: Improved Prediction of Clinical Outcome With the Use of Global Strain and Mechanical Dispersion in Patients With Myocardial Infarction and Heart Failure
Brief Title: Global Strain and Mechanical Dispersion May Predict Death and Ventricular Arrhythmias Better Than Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Thor Edvardsen, Professor, Chief department of Cardiology Oslo university hospital, Oslo University Hospital
Other Study IDs: 2013/573/REK sør-øst
Record Dates: First submitted 2014-08-22; First posted 2014-11-10 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Left Ventricular Function Systolic Dysfunction
Keywords: Ejection fraction, Global Strain, Mechanical dispersion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate if global strain and mechanical dispersion may predict death and ventricular arrhythmias better than ejection fraction(EF) in patients with myocardial infarction and heart failure regardless of cause.

DETAILED DESCRIPTION:
1. The main aim of this study is to investigate if global strain and mechanical dispersion may predict death and ventricular arrhythmias better than left ventricular ejection fraction in patients with myocardial infarction and heart failure.
2. In patients who receive internal cardioverter defibrillator(ICD) the main aim is to investigate if mechanical dispersion may predict ventricular arrhythmias better than EF.

3) No interventions,only evaluation of the measurements obtained with transthoracic echocardiography.

4) Follow up for 3 years, extended from 3 to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients with

  1. myocardial infarction
  2. heart failure( defined as heart failure symptoms: reduced left ventricular function/ and or heart failure signs on chest x ray.
  3. planned for primary prophylactic ICD
* over 18 years of age
* Informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myocardial infarction, heart failure and patients planned for primary prophylactic ICD. Echocardiography is performed at inclusion. Comparism of the ability of left ventricular ejection fraction, global strain and mechanical dispersion to predict clinical outcome in patients with these conditions.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmia and death after acute myocardial infarction or heart failure. | 5 years or more
  Arrhythmic events during follow-up are defined as documented sustained ventricular tachycardia, ventricular fibrillation, and SCD. Survival is assessed by medical charts if patients are within the uptake area of the hospital and by the Norwegian death registry Folkeregisteret.

CONTACTS AND LOCATIONS:
Overall Officials: Thor Edvardsen, MD, PHD, Study Director — Oslo University Hospital
Locations (8):
- Vseobecna fakultni nemocnice Praha/ Prague General hospital, Prague, Czechia
- Norway (7):
  - Sørlandet sykehus HF, Arendal, Agder
  - Vestre Viken HF, Drammen
  - Sørlandet sykehus Kristiansand, Kristiansand
  - Oslo university hospital, Oslo
  - Sykehuset Telemark HF, Skien
  - Stavanger universitetssjukehus, Stavanger
  - Universitetssykehuset Nord Norge, Tromsø, Tromsø

IPD SHARING:
Plan to Share IPD: Undecided